CLINICAL TRIAL: NCT02373397
Title: Cacicol20® in Corneal Wound Healing and Nerve Regeneration After Phototherapeutic Keratectomy of the Anterior Cornea: A Randomized Double-Blinded Placebo-Controlled Study
Brief Title: Cacicol20® in Corneal Wound Healing and Nerve Regeneration After Phototherapeutic Keratectomy
Acronym: CACICOL-PTK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to poor patient recruitment
Sponsor: Neil Lagali (Other)
Collaborators: Region Östergötland (Other); Linkoeping University (Other Government); Sahlgrenska University Hospital (Other); Laboratoires Thea (Industry)
Responsible Party: Sponsor-Investigator, Neil Lagali, Associate Professor, Region Östergötland
Organization: Region Östergötland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2014/465-31
Record Dates: First submitted 2015-02-16; First posted 2015-02-27 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Corneal Dystrophy, Epithelial Basement Membrane; Epithelial Recurrent Erosion Dystrophy; Corneal Erosions
Keywords: Wound healing; nerve regeneration; re-epithelialization; corneal epithelium; laser corneal surgery
MeSH Terms: conditions — Corneal dystrophy, epithelial basement membrane; Epithelial Recurrent Erosion Dystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cacicol20 (Experimental): Instillation of Cacicol20 eye drops after laser corneal surgery. 3 eye drops total, to be given once immediately after surgery, once 2 days after surgery, and a final time 4 days after surgery.
  Interventions: Device: Cacicol20
- Placebo (Placebo Comparator): Instillation of placebo eye drops (vehicle missing the active ingredient) after laser corneal surgery. 3 eye drops total, to be given once immediately after surgery, once 2 days after surgery, and a final time 4 days after surgery.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Cacicol20 — Investigational device, regenerating agent, single-use doses, topical eye drops. Indicated for corneal wound healing.
  Other Names: RGTA; Cacicol; RGTA OTR 4120
  Arms: Cacicol20
Device: Placebo — Vehicle only in identical packaging, with identical dosage and administration route.
  Arms: Placebo

SUMMARY:
The objective of this clinical study is to test the efficacy of CACICOL20® (RGTA OTR 4120) in improving wound healing and nerve regeneration in the anterior cornea, in a patient population undergoing therapeutic laser treatment for corneal dystrophy or recurrent corneal erosions.

DETAILED DESCRIPTION:
Patients undergoing various surgical treatments of the cornea often suffer from a neural deficit, due to nerves being severed or removed completely during surgery. This can result in pain, impaired epithelial wound healing, reduced tear production, symptoms of dry eye, and loss of ocular surface sensitivity/blink reflex. In addition, surgical wound healing can be accompanied by undesirable formation of scar tissue, which can limit postoperative visual acuity. The investigators' prior clinical experience with patients having undergone surgery of the anterior cornea is that neural recovery is slow and incomplete, while in certain situations scar tissue can form and limit the visual recovery.

In this context, CACICOL20®, a regenerative agent approved for use in healing corneal wounds, presents an interesting opportunity for improving postoperative corneal nerve regeneration and a potentially more rapid restoration of the extracellular matrix environment postoperatively, which can lead to improved neural and visual outcomes.

The investigators will therefore evaluate the efficacy of CACICOL20® in a randomized, double-blinded clinical study, to evaluate its ability to promote corneal nerve regeneration, epithelial wound healing, and ocular surface recovery postoperatively.

Upon inclusion and signing of informed consent, patients undergo preoperative examination. Upon satisfying study criteria, patients are randomized to either treatment or placebo group. Group identity is masked to subjects and to investigators (double-blind). Subjects then undergo therapeutic laser treatment of the cornea in a single clinic, followed by instillation of treatment or placebo in the form of 3 eye drops total (to be given once immediately after surgery, once 2 days after surgery, and a final time 4 days after surgery).

Postoperative eye examinations are conducted on days 2 and 7 and at month 6 and 12. Examinations include clinical measurement of various eye and corneal wound healing parameters.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent,
* Male or female aged ≥ 18 years,
* Patient with recurrent erosions or epithelial dystrophies indicated for treatment by phototherapeutic keratectomy of the anterior cornea

Exclusion Criteria:

* In the affected eye: prior corneal surgery
* In either eye: active ocular infection, glaucoma, or ocular hypertension
* General history judged by the investigator to be incompatible with the study (life-threatening patient condition).
* Known allergic hypersensitivity history to Poly(carboxyMethylGlucoseSulfate) or dextran.
* Inability of patient to understand the study procedures and thus inability to give informed consent.
* Participation in another clinical study within the last 3 months.
* Already included once in this study (can only be included for one treated eye)

Specific exclusion criteria for women

* Known pregnancy (if uncertain pregnancy test will be performed)
* Lactation
* Women of childbearing potential without an effective method of contraception (oral contraceptive, intra-uterine device, subcutaneous contraceptive implant, vaginal ring) or women not hysterectomised, post-menopausal or surgically sterilized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage recovery in subbasal nerve density. | 12 months postoperative
  Degree of corneal subbasal nerve regeneration at one year postoperative, compared to preoperative level, as measured by clinical laser-scanning in vivo confocal microscopy.

SECONDARY OUTCOMES:
Percentage recovery in subbasal nerve density. | 6 months postoperative
  Degree of corneal subbasal nerve regeneration at 6 months postoperative, compared to preoperative level, as measured by clinical laser-scanning in vivo confocal microscopy.
Percentage of epithelial wound closure. | 2 and 7 days postoperative.
  A drop of sodium fluorescein liquid is applied to the cornea, and a digital photograph is taken at high magnification with a clinical slit lamp biomicroscope, using a blue illumination lamp. Area of open wound is measured from photographs and expressed as a percentage of the total treated area.
Postoperative pain score on the Visual Analog Scale. | Postoperative day 2, 7, month 6, 12
  Patient self-assessment using the subjective VAS scale (100 point scale).
Corneal haze level. | Postoperative month 6, 12
  Corneal haze measured microscopically by clinical in vivo confocal microscopy using a semi-quantitative grading scale.
Number of postoperative recurrences of erosions. | Postoperative month 12.
  As reported by the patient.
Ocular surface sensitivity measured by Cochet-Bonnet esthesiometry. | Postoperative month 6, 12
  Central corneal mechanical touch sensitivity in mm measured by Cochet-Bonnet esthesiometry.
Tear production level | Postoperative day 7, month 6, 12
  Tear production level (in mm) measured by the Schirmer test without anesthetic.
Tear quality | Postoperative day 7, month 6, 12
  Tear break up time (in seconds) timed by slit lamp biomicroscopic observation after instillation of sodium fluorescein and induction of blinking.
Improvement in visual acuity | Postoperative day 7, month 6, 12
  Distance corrected visual acuity improvement measured in Snellen lines gained/lost relative to preoperative level.
Sub basal nerve density measured by clinical in vivo confocal microscopy | Postoperative 6 and 12 months
  Sub basal nerve density level measured by clinical in vivo confocal microscopy.
Epithelial cell density measured by clinical in vivo confocal microscopy | Postoperative 12 months
  Epithelial wing cell density measured by clinical in vivo confocal microscopy.

OTHER OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability. | From operation day until 12 months postoperative.
  Defined as reactions or complications beyond those normally expected after laser corneal surgery. Assessed by the investigator.
Number of patients using supplementary eye treatments. | Operation day until 12 months postoperative.
  Use of any supplementary eye treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Jarkman, MD PhD, Study Chair — Region Östergötland
Locations (2):
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Sahlgrenska University Hospital, Mölndal

REFERENCES:
- [Background] Meddahi A, Alexakis C, Papy D, Caruelle JP, Barritault D. Heparin-like polymer improved healing of gastric and colic ulceration. J Biomed Mater Res. 2002 Jun 5;60(3):497-501. doi: 10.1002/jbm.1293. PMID 11920675
- [Background] Chebbi CK, Kichenin K, Amar N, Nourry H, Warnet JM, Barritault D, Baudouin C. [Pilot study of a new matrix therapy agent (RGTA OTR4120) in treatment-resistant corneal ulcers and corneal dystrophy]. J Fr Ophtalmol. 2008 May;31(5):465-71. doi: 10.1016/s0181-5512(08)72462-8. French. PMID 18641578
- [Background] Lagali N, Germundsson J, Fagerholm P. The role of Bowman's layer in corneal regeneration after phototherapeutic keratectomy: a prospective study using in vivo confocal microscopy. Invest Ophthalmol Vis Sci. 2009 Sep;50(9):4192-8. doi: 10.1167/iovs.09-3781. Epub 2009 Apr 30. PMID 19407024
- [Background] Germundsson J, Lagali N. Pathologically reduced subbasal nerve density in epithelial basement membrane dystrophy is unaltered by phototherapeutic keratectomy treatment. Invest Ophthalmol Vis Sci. 2014 Mar 25;55(3):1835-41. doi: 10.1167/iovs.13-12533. PMID 24569577
- [Background] Cejkova J, Olmiere C, Cejka C, Trosan P, Holan V. The healing of alkali-injured cornea is stimulated by a novel matrix regenerating agent (RGTA, CACICOL20): a biopolymer mimicking heparan sulfates reducing proteolytic, oxidative and nitrosative damage. Histol Histopathol. 2014 Apr;29(4):457-78. doi: 10.14670/HH-29.10.457. Epub 2013 Oct 9. PMID 24105332
- [Background] De Monchy I, Labbe A, Pogorzalek N, Gendron G, M'Garrech M, Kaswin G, Labetoulle M. [Management of herpes zoster neurotrophic ulcer using a new matrix therapy agent (RGTA): A case report]. J Fr Ophtalmol. 2012 Mar;35(3):187.e1-6. doi: 10.1016/j.jfo.2011.09.002. Epub 2011 Oct 19. French. PMID 22015067
- [Background] Kymionis GD, Liakopoulos DA, Grentzelos MA, Diakonis VF, Klados NE, Tsoulnaras KI, Tsilimbaris MK, Pallikaris IG. Combined topical application of a regenerative agent with a bandage contact lens for the treatment of persistent epithelial defects. Cornea. 2014 Aug;33(8):868-72. doi: 10.1097/ICO.0000000000000169. PMID 24937169